CLINICAL TRIAL: NCT06598475
Title: Investigating Facilitator-driven, Multi-level Implementation Strategies in Federally Qualified Health Centers to Improve Provider Recommendation and HPV Vaccination Rates Among Latino/a Adolescents
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Daisy Y. Morales Campos, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: HSC-SPH-24-0335
Record Dates: First submitted 2024-09-13; First posted 2024-09-19 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Human Papillomavirus Infection
Keywords: HPV vaccination
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Intervention Model Description: This is a stepwise cluster randomized control design study. There will be 3 clusters (FQHC's) having 3 practices each
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Step 1 (3 clinics)-15 months control then 30 months intervention (Experimental)
  Interventions: Other: Facilitator-driven provider- and practice-level implementation strategies for influencing provider recommendations and practice-level HPV vaccination rates
- Step 2 (3 clinics)-21 months control then 24 months intervention (Experimental)
  Interventions: Other: Facilitator-driven provider- and practice-level implementation strategies for influencing provider recommendations and practice-level HPV vaccination rates
- Step 3 (3 clinics)-27 months control then 18 months intervention (Experimental)
  Interventions: Other: Facilitator-driven provider- and practice-level implementation strategies for influencing provider recommendations and practice-level HPV vaccination rates

INTERVENTIONS:
Other: Facilitator-driven provider- and practice-level implementation strategies for influencing provider recommendations and practice-level HPV vaccination rates — The practice facilitator (UTHealth research staff) will implement the following 4 strategies with providers and immunization navigators at each practice:
  * Facilitator-driven provider education: The practice facilitator will conduct one provider education module (5 total modules) over three months with health care providers using a booklet and resource binder.
  * Facilitator-driven clinical practice plan: The practice facilitator will assist the implementation team in creating their clinical practice in two additional modules and encourage providers to identify strategies to increase HPV vaccination.
  * Training and education for staff (Immunization Navigators): The facilitator will train immunization navigators to implement the plan, and practice immunization navigators will implement the plan.
  * Technical assistance plus assessment and feedback: During implementation of the plan, the facilitator will provide technical assistance, ongoing assessment and feedback, and booster trainings.

SUMMARY:
The purpose of this study is to determine the provider- and practice-level characteristics that influence the impact of implementation strategies guided by practice facilitation in each clinical practice, to test whether the facilitator-driven provider- and practice-level implementation strategies increase provider recommendations and Human Papilloma Virus (HPV) vaccination rates and to evaluate implementation and future sustainability of the facilitator-driven implementation strategies across nine clinical practice sites

ELIGIBILITY:
Inclusion Criteria:

* FQHC's with less than 60% HPV vaccine initiation rate for 11-12 year old adolescents overall at their practice sites
* FQHC's that have family medicine and/or pediatric practices
* a total adolescent patient population at least 50% Latino
* be willing for Health Care Provider (HCP) and staff members to receive education, training, and support; complete standardized measurement, and agree to randomization.
* Providers, aged 18 and over, employed at each FQHC (4 staff per practice)
* Staff, aged 18 and over, employed at each FQHC (5 staff per practice)
* Implementation team members (i.e., administrative designee, health care providers, immunization navigators, and other staff), aged 18 and over, employed at each FQHC (4 members per practice)
* Parents (aged 18 and over) of patients ages 11-17 seeking care at each FQHC (25 per practice).

Exclusion Criteria:

-FQHCs that participated in the pilot study were excluded.

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2142 (Estimated)
Dates: Start 2025-03-13 (Actual); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of vaccine-eligible males and females at each clinic who received the first valid dose of the HPV vaccine series before their 13th birthday. | From baseline to end of study ( about 60 months from baseline)
Percentage of vaccine-eligible males and females at each clinic who received the second valid dose of the HPV vaccine series 6-12 months after their first dose and before their 13th birthday. | From baseline to end of study ( about 60 months from baseline)

SECONDARY OUTCOMES:
Percentage of vaccine-eligible males and females at each clinic who received the first valid dose of the HPV vaccine series before their 18th birthday. | From baseline to end of study ( about 60 months from baseline)
Percentage of vaccine-eligible 13-14 y/o males and females at each clinic who received the second valid dose of the HPV vaccine series 6-12 months after first dose and before their 15th birthday | From baseline to end of study ( about 60 months from baseline)
Percentage of vaccine-eligible 15-17 y/o males and females at each clinic who received the second valid dose of the HPV vaccine series 2 months after first dose and before their 18th birthday | From baseline to end of study ( about 60 months from baseline)
Percentage of vaccine-eligible 15-17 y/o males and females at each clinic who received the third valid dose of the HPV vaccine series 4 months after second dose and before their 18th birthday. | From baseline to end of study ( about 60 months from baseline)
Percentage of non-well visits in which HPV vaccine was not administered, among all visits for active vaccine-eligible patients ages 11-17 by clinic | From baseline to end of study ( about 60 months from baseline)
Percentage of males and females at each clinic who received Tdap and MenACWY at age 11 as a requirement to attend 7th grade in Texas. | From baseline to end of study ( about 60 months from baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Daisy Y Morales Campos, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Morales-Campos DY, Adsul P, Liang Y, Donovan E, Moczygemba LR, Kahn JA. Trusted health system implementation strategies to increase vaccination (TRUE SYNERGI): a stepped-wedge cluster randomized trial to reduce HPV-related cancers. BMC Public Health. 2025 Apr 9;25(1):1331. doi: 10.1186/s12889-025-22273-7. PMID 40205591